CLINICAL TRIAL: NCT03373500
Title: A Randomised Controlled Trial of the Effect of Dietary Salt Reduction on Blood Pressure and Other Cardiovascular Parameters in Kidney Transplant Recipients
Brief Title: Effect of Dietary Salt Reduction on Blood Pressure in Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Epsom and St Helier University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002S/2016/REN
Record Dates: First submitted 2017-11-29; First posted 2017-12-14 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Blood Pressure; Hypertension; Kidney Transplant; Complications; Dietary Modification
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Single centre, randomised controlled parallel study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Salt Diet (Experimental): Dietary salt reduction: Patients will be given intensive dietary advice to achieve a low salt diet, targeting a dietary salt intake of less than 5g per day (80 mmol/day).
  Interventions: Other: Dietary salt reduction
- Standard Treatment (No Intervention): Patients will be instructed to continue with their usual diet, therefore no advice will be given about salt reduction.

INTERVENTIONS:
Other: Dietary salt reduction — Patients will be given intensive dietary advice to achieve a low salt diet, targeting a dietary salt intake of less than 5g per day (80 mmol/day).
  Arms: Low Salt Diet

SUMMARY:
Cardiovascular morbidity and mortality is increased in kidney transplant patients. High blood pressure (BP) contributes significantly to this risk and is also associated with shortened allograft survival. Salt reduction lowers BP in the general population and there is emerging data that salt reduction also effectively lowers BP in chronic kidney disease (CKD). Kidney transplant patients, by definition have CKD, but they differ fundamentally from the general CKD population in that they are on medications which can predispose to high blood pressure, their kidneys are denervated, and they often have reasonable excretory kidney function.

The proposed study will be an eight-week randomised, controlled trial assessing the effect of intensive dietary salt advice on cardiovascular risk factors in kidney transplant patients. The primary outcome is office BP readings, with the effect on 24-hour ambulatory blood pressure, proteinuria, arterial stiffness and endothelial function being studied as secondary outcomes.

DETAILED DESCRIPTION:
Our hypothesis is that lower salt intake will reduce BP in patients with a kidney transplant. We propose that this will translate into better CV and renal protection via reductions in proteinuria, endothelial dysfunction and arterial stiffness.

The primary aim of the study is to examine the impact of reduced dietary salt intake on blood pressure (BP) in kidney transplant patients. Secondary aims include examination of the effect of salt reduction on ambulatory blood pressure parameters, markers of proteinuria, endothelial and metabolic dysfunction, arterial stiffness and renal fibrosis.

The study will be a single centre, randomised controlled parallel study. Individuals aged 18 years old and above will be recruited from the kidney transplant population of the South West Thames Renal Unit. Patients who have received a kidney transplant ≥ 6 months previously who have a BP >130 mm Hg systolic and/or >80 mm Hg diastolic, or are receiving treatment for hypertension will be included.

Informed consent will be obtained from all study participants and each patient will be given a patient information sheet. At the beginning of the 2-week run-in period individuals will be assessed for eligibility with office BP readings and a 24hr urine collection. Baseline measurements will be taken whilst participants are on their usual diet. All measurements will be performed at baseline, after a 2-week run in period, and at the end of the 8-week study period.

After baseline measurements are taken at the end of the 2-week run in period, participants will be randomised to either the low salt arm or the standard treatment arm using computer-generated randomisation. Patients will be asked to bring in a food diary from the weekend and two week days so that dietary advice can be tailored to the individual. Patients allocated to the low salt diet group will be advised by a doctor to achieve a dietary salt intake of less than 5g per day (80mmol/day). The control group will be instructed to continue with their usual diet, therefore no advice will be given about salt reduction, but otherwise the groups will follow an identical trial protocol.

In addition patients will be seen at week two for a BP reading and a 24hr urine collection, and at week four for a BP reading, 24hr urine collection and measurement of renal profile (Not fasted). Advice will be reinforced at each visit and through telephone for the duration of the study. Antihypertensive treatment will remain unchanged throughout the study apart from two caveats: If BP rises >160/100 then a further antihypertensive will be added at the attending physicians discretion; If BP drops <90/60 and/or symptomatic hypotension, antihypertensive treatment will be withdrawn at the attending physicians discretion, with further investigation as necessary.

Blood pressure will be measured using a validated oscillometric technique, in the sitting position, after 5 to 10 minutes rest and using the same arm throughout the study. Three readings at 1-2 minute intervals will be taken and the mean of the last 2 readings will be used for analysis. Twenty-four hour ambulatory BP monitoring will be performed using a validated oscillometric system. Two 24-hour urine collections for the measurement of sodium, potassium, urea, and creatinine, will be performed at baseline and at the end of the 8-week study period. Blood and urine samples will be taken after an overnight fast (8 - 14 hr) at baseline and then end of the study for measurement of routine biochemistry, plasma renin activity, aldosterone, urinary protein creatinine ratio and urinary albumin creatinine ratio. Blood and urine samples will be taken at baseline and the end of study assessment to look at markers of endothelial function and novel markers of renal dysfunction and fibrosis. These will include EDA+Fibronectin, transforming growth factor-β (TGF-β) and connective tissue growth factor (CTGF).

Endothelial function and arterial stiffness will be assessed by digital volume pulse analysis (DVP) using a high-fidelity photo-plethysmography (PulseTrace1000, MicroMedical Ltd, Rochester, Kent, U.K). Changes in the reflective index (RI) following salbutamol administration are measured as a test of endothelial vasodilatory function and changes following glyceroltrinitrate (GTN) are measured as a test of endothelium independent vasodilation. Baseline measurements are taken in triplicate at 5 min intervals after subjects lay quietly for 20 min. Sublingual GTN 500mcg (Alpharma, Barnstable, Devon, U.K.) is administered for 3 min and recordings are made at 3, 5, 10, 15 and 20 min. Following a rest of 10 min, albuterol 400mcg (salbutamol, Baker Norton, London, U.K.) is administered via a spacer device and recordings are repeated at 5, 10 and 15 min. This technique is validated for measuring endothelial function with reproducibility for change in reflective index following albuterol (∆RIAlb) of -1.9±4.9% and following GTN (∆RIGTN) of -2.2±5.4%.

To measure arterial stiffness using DVP, the systolic peak and inflection point are obtained by analysing the first derivative of DVP waveforms. The time between first systolic peak and the inflection point in the waveforms (∆TDVP) is determined. The DVP-derived stiffness index (SIDVP) is calculated by the following equation: body height /∆TDVP.

A single trained operator will perform all vascular measurements after an overnight fast in a quiet temperature controlled room.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a kidney transplant ≥ 6 months previously who have a BP >130 mm Hg systolic and/or >80 mm Hg diastolic, or are receiving treatment for hypertension.

Exclusion Criteria:

* BP < 120/80 on blood pressure treatment
* BP >160/100
* Variation in Creatinine >20% over preceding 2 months
* Secondary hypertension due to a cause other than CKD
* Heart failure (LVEF <30% or NYHA class II - IV)
* Myocardial Infarction within 6 months
* Stroke within 6 months
* Current diagnosis of cancer
* Liver disease
* Bilateral arterio-venous fistulae
* Evidence of significant active infection
* Females who are pregnant or breastfeeding
* Hyponatremia (Na <130mmol/L) or Hypernatremia (Na >150mmol/L)
* Histologically confirmed episode of rejection within 6 months
* Steroids dose change in preceding 2 months
* Patients who are not able to give full informed consent
* Initial 24hr urinary sodium <80mmol/24hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Office systolic and diastolic BP readings | 9 months
  Systoli and diastolic BP measurements in mmHg

SECONDARY OUTCOMES:
Ambulatory BP monitoring | 9 months
  Total 24 hour average systolic and diastolic BP measurements in mmHg
Endothelial function, measured by digital pulse wave analysis (DVP) | 9 months
  Endothelial dependent function will be calculated as the difference between the mean measurements of the baseline reflective index (RI) measurements and the RI following Salbutamol inhalation and endothelium independent function is calculated as the difference between the mean of the baseline RI measurements and the RI following administration of glyceroltrinitrate (GTN)
Arterial stiffness, measured by digital pulse wave analysis (DVP) | 9 months
  The systolic peak and inflection point are obtained by analysing the first derivative of DVP waveforms. The time between first systolic peak and the inflection point in the waveforms (∆TDVP) is determined. The DVP-derived stiffness index (SIDVP) is calculated by the following equation: body height /∆TDVP.
Proteinuria | 9 months
  Urinary protein creatinine ratio in g/mol and albumin creatinine ratio in g/mol
Biomarkers of fibrosis | 9 months
  TGF-β1, 2 & 3 will be measured on a multiplex platform using a Bioplex analyser. CTGF & EDA+Fibronectin levels will be assesed by semi-quantitative Western Blotting, which will identify full length proteins and also biologically relevant fragments and isoforms. EDA+Fibronectin will be compared to total Fibronectin using an adaptation of a commercial ELISA. Levels of CTGF in the plasma will also be measured. These urinary and plasma biomarkers can then be correlated with the 48hr urinary sodium excretion performed at the beginning and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Swift, MBBS, Principal Investigator — Epsom and St Helier University Hospitals NHS Trust
Locations (1):
- Epsom and St Helier University Hospitals NHS Trust, Carshalton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803